CLINICAL TRIAL: NCT06123923
Title: Contemporary Patterns and Underlying Causes of Vitrectomy in Pediatric and Adolescent Patients: A Nationwide, Population-Based Analysis
Brief Title: Trends of Vitreoretinal Surgery in Children
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kunho Bae, MD, Seoul National University Hospital
Other Study IDs: IRB No. 2022-07-010
Record Dates: First submitted 2023-11-03; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Vitreoretinal Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention, just retrospective observation

SUMMARY:
Purpose: We determined the incidence, etiology, and longitudinal trends of vitreoretinal diseases necessitating pars plana vitrectomy (PPV) in the pediatric and adolescent population.

Design: This was a nationwide, population-based cohort study, utilizing data from the Korean National Health Claims database spanning from 2009 to 2020.

Given the retrospective design of the study and the anonymized nature of the data, the requirement for informed consent was waived.

Methods: All pediatric and adolescent patients (under 20 years of age) who underwent PPV across the Korean population were included. The cumulative incidence of PPV was estimated from 2009 to 2020, with 2009 to 2011 as the washout period. The annual trends of PPV incidence, the proportion of each etiology, and comorbidity were estimated based on sex and specific age groups.

ELIGIBILITY:
Inclusion Criteria:

* We included all pediatric and adolescent patients who underwent complete PPV (registered under code S5121) during the study period from January 2009 to December 2020, and who were continuously enrolled in a medical plan, in our estimates.

Ages: 0 Years to 19 Years | Sex: All
Age Groups: Child, Adult
Study Population: all pediatric and adolescent subjects under 20 years of age in Korean population
Sampling Method: Probability Sample
Enrollment: 3509 (Actual)
Dates: Start 2022-10-16 (Actual); Primary Completion 2022-12-17 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
number of vitreoretinal surgery | 2009-2020
  vitreoretinal surgeries that had already performed during the retrospective study period

CONTACTS AND LOCATIONS:
Overall Officials: Kunho Bae, MD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided